CLINICAL TRIAL: NCT04339361
Title: Comparative Safety and Efficacy of Lidocaine Spray Versus Vaginal Dinoprostone in Relieving Pain During Levonorgestrel IUD Insertion
Brief Title: Comparative Efficacy of Lidocaine Spray Versus Vaginal Dinoprostone in IUD Insertion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: lidocaine spray IUD
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Contraception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lidocaine spray (Experimental): four puffs (50ml, 10 mg/puff) of lidocaine spray will be applied to the cervical canal and cervix before tenaculum placement plus vaginal placebo will be given 3 hours before IUD insertion
  Interventions: Drug: lidocaine spray
- vaginal dinoprostone (Active Comparator): vaginal dinoprostone 3 mg will be given 3 hours before IUD insertion plus four puffs of saline spray will be applied to the cervical canal and cervix before tenaculum placement
  Interventions: Drug: vaginal dinoprostone
- placebo (Placebo Comparator): vaginal placebo will be given 3 hours before IUD insertion plus four puffs of saline spray will be applied to the cervical canal and cervix before tenaculum placement
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lidocaine spray — four puffs (50 ml, 10 mg/puff) of lidocaine spray before tenaculum placement plus vaginal placebo 3 hours before IUD insertion
  Arms: lidocaine spray
Drug: vaginal dinoprostone — vaginal dinoprostone 3 mg will be given 3 hours before IUD insertion plus four puffs of saline spray before tenaculum placement
  Arms: vaginal dinoprostone
Drug: placebo — vaginal placebo will be given 3 hours before IUD insertion plus four puffs of saline spray before tenaculum placement
  Arms: placebo

SUMMARY:
the aim of this study is to compare the safety and Efficacy of Lidocaine Spray Versus Vaginal dinoprostone in relieving pain during levonorgestrel IUD Insertion in nulliparous women

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women requesting levonorgestrel IUD insertion

Exclusion Criteria:

* multiparous women, allergy or contraindication to study drugs or contraindications to LNG-IUD insertion

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2020-04-25 (Estimated); Primary Completion 2020-08-10 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
pain during IUD insertion | 2 minutes
  pain during IUD insertion assessed by 10 cm visual analog scale where 0 denotes no pain and 10 denotes the worst pain imaginable

SECONDARY OUTCOMES:
insertion duration | 5 minutes
  duration of LNG-IUD insertion from speculum in to speculum out